CLINICAL TRIAL: NCT03842215
Title: Development and Clinical Applications of a Smart Physical Examination System for the Health Management in Elderly
Brief Title: A Smart Physical Examination System for the Health Management in Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CCH-181211
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Physical Activity
Keywords: smart physical examination system; health management; elderly
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- silver hair people: Exam subject's physical function by a smart physical exam
  Interventions: Device: smart physical exam

INTERVENTIONS:
Device: smart physical exam — Use smart physical exam to collect functional performance

SUMMARY:
The object of this study is to develop a smart physical examination system targeted on the unmet need of the elderly.Furthermore,the ultimate goal is to realize a commercial product aiming at the silver hair market with functional advantages to meet the unmet needs of health management in elderly.

DETAILED DESCRIPTION:
Aging usually results in a decline of motor function. However, elderly tends to refuse the regular health examination because of travel issues or lack of self-health awareness. Examination unit also has difficulty to intensively track and instantly feedback the health status of elderly due to insufficient manpower. If elderly goes to the hospital only when the health problem is getting worse, his/her health is often irreversible and the cost of medical care would be increased. It is therefore an essential issue for the early detection of functional changes in elderly to prevent the deterioration of the health and function. Currently, the telemedicine cares provided by hospitals are not universal due to the out-of-date legislation and non-successful business model. The wearing and operation issues of the wearable devices used for health management are still a gap affecting the acceptance of elderly. Accordingly, the objective of this project is to develop a handy and easy-to-use smart physical examination system targeted on the unmet need of the elderly. With the use of motion-sensing and big data analysis technology, the non-contact professional and intelligent assessment could simplify the general health checkup procedures to promote the health management and to reduce the manpower cost of health care. Following the principle of commercialization, this project aims at working out the product prototype, finalize the assessment tools/algorithm, and put it into the clinical trials. The project research team comprising the physicians, therapists, hardware and software systems engineering experts, with the early manufacturing involvement from the industry partner. The team members will work closely to solve the clinical, engineering, and market demand issues during the development process. The project will build a platform to deepen the bilateral understanding and research cooperation to solve the aging society problem. The ultimate goal is to realize a commercial product aiming at the silver hair market with functional advantages to meet the unmet needs of health management in elderly.

ELIGIBILITY:
Inclusion Criteria:

1.55-85 years old 2.people who can do movement by 3.people who can walk >10m independently.

Exclusion Criteria:

1. people who implant cardiac rhythm, have cardiac arrhythmia,tumor,infection,or any other internal disease.
2. people who have visual disturbance (Corrected vision<4.0 or any ophthalmic diseases caused bad eyesight),hearing loss,movement disorder.
3. people who can't stand stably.
4. people who can't fill out a questionnaire independently.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling people who are recruited from the local community, hospital, club.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Single Leg Balance Test | Test once while subject is recruited.
  Remove the shoes and stand on the floor. Stand on one leg for 60 seconds and record the duration (seconds) that subject keeps one leg stand.
  The test is stopped
  1. if the legs touch each other,
  2. if the weight-bearing foot moves on the floor,
  3. if the non-weight bearing foot touches the floor
  4. if the hands are removed from the waist.
Functional Reach Test | Test once while subject is recruited.
  Position the patient close to the wall. The patient is instructed to stand with feet shoulder distance apart then make a fist and raise the arm up so that it's parallel to the floor.
  At this time, the practitioner takes an initial reading on the yardstick, usually spotting the knuckle of the third metacarpal.
  The patient is instructed to reach forward along the yardstick without moving the feet, the hand should remain in a fist.
  The practitioner takes a reading on the yardstick of the farthest reach (cm) attained by the patient without taking a step.
Chair Sit and Reach Test | Test once while subject is recruited.
  The subject sits on the edge of a chair. One foot must remain flat on the floor. The other leg is extended forward with the knee straight, heel on the floor, and ankle bent at 90°. Place one hand on top of the other with tips of the middle fingers even. Instruct the subject to Inhale, and then as they exhale, reach forward toward the toes by bending at the hip. Keep the back straight and head up.
  Keep the knee straight, and hold the reach for 2 seconds. The distance is measured between the tip of the fingertips and the toes. If the fingertips touch the toes then the score is zero. If they do not touch, measure the distance between the fingers and the toes (a negative score), if they overlap, measured by how much (a positive score). Perform two trials.
  The score is recorded to the nearest 1/2 inch or 1 cm as the distance reached, either a negative or positive score. Record which leg was used for measurement.
2 minute step | Test once while subject is recruited.
  The subject stands up straight next to the wall while a mark is placed on the wall at the level corresponding to midway between the patella (knee cap) and iliac crest (top of the hip bone). The subject then marches in place for two minutes, lifting the knees to the height of the mark on the wall. Resting is allowed, and holding onto the wall or a stable chair is allowed. Stop after two minutes of stepping, and measure the heart rate (beats/min).
Arm Curl Test | Test once while subject is recruited.
  The aim of this test is to do as many arm curls as possible in 30 seconds. This test is conducted on the dominant arm side. The subject sits on the chair, holding the weight in the hand using a suitcase grip with the arm in a vertically down position beside the chair. Brace the upper arm against the body so that only the lower arm is moving. Curl the arm up through a full range of motion, gradually turning the palm up (flexion with supination). As the arm is lowered through the full range of motion, gradually return to the starting position. The arm must be fully bent and then fully straightened at the elbow. Repeat this action as many times as possible within 30 seconds.
  The repetitions of arm curl are recorded.
30-sec sit -to-stand | Test once while subject is recruited.
  Use 30-Second sit to stand to test leg strength and endurance.
  1. Sit in the middle of the chair.
  2. Place your hands on the opposite shoulder crossed, at the wrists.
  3. Keep your feet flat on the floor.
  4. Keep your back straight, and keep your arms against your chest.
  5. On "Go," rise to a full standing position, then sit back down again.
  6. Repeat this for 30 seconds.
  7. Record the repetitions is performed.
Euro QOL-5D | Test once while subject is recruited.
  The Euro QOL-5D (EQ-5D) comprises five questions on mobility, self-care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem).
  A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores.
  The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analog scale (VAS) to indicate the general health status with 100 indicating the best health status.
International Physical Activity Questionnaire (IPAQ) | Test once while subject is recruited.
  IPAQ comprises a set of 4 questionnaires and will ask about the time the subject spent being physically active in the last 7 days.
  Three levels (categories) of physical activity are proposed:
  Category 1: Low Those individuals who not meet criteria for categories 2 or 3 are considered low/inactive.
  Category 2: Moderate
  Any one of the following 3 criteria:
  * 3 or more days of vigorous activity of at least 20 minutes per day OR
  * 5 or more days of moderate-intensity activity or walking of at least 30 minutes per day OR
  * 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 MET-min/week.
  Category 3: High
  Any one of the following 2 criteria:
  * Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/week OR
  * 7 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 3000 MET-minutes/week

CONTACTS AND LOCATIONS:
Overall Officials: TaSen Wei, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No
only for search

REFERENCES:
- [Background] Arias-Palencia NM, Solera-Martinez M, Gracia-Marco L, Silva P, Martinez-Vizcaino V, Canete-Garcia-Prieto J, Sanchez-Lopez M. Levels and Patterns of Objectively Assessed Physical Activity and Compliance with Different Public Health Guidelines in University Students. PLoS One. 2015 Nov 4;10(11):e0141977. doi: 10.1371/journal.pone.0141977. eCollection 2015. PMID 26536605
- [Background] Choi JS, Kang DW, Seo JW, Kim DH, Yang ST, Tack GR. The development and evaluation of a program for leg-strengthening exercises and balance assessment using Kinect. J Phys Ther Sci. 2016 Jan;28(1):33-7. doi: 10.1589/jpts.28.33. Epub 2016 Jan 30. PMID 26957724
- [Background] Franz-Ritscherle A, Lange DE. [Effectiveness of various audiovisual technics to improve oral hygiene behavior]. Dtsch Zahnarztl Z. 1983 Sep;38(9):811-5. No abstract available. German. PMID 6196174
- [Background] Handrigan GA, Maltais N, Gagne M, Lamontagne P, Hamel D, Teasdale N, Hue O, Corbeil P, Brown JP, Jean S. Sex-specific association between obesity and self-reported falls and injuries among community-dwelling Canadians aged 65 years and older. Osteoporos Int. 2017 Feb;28(2):483-494. doi: 10.1007/s00198-016-3745-x. Epub 2016 Aug 25. PMID 27562568
- [Background] Jorgensen MG. Assessment of postural balance in community-dwelling older adults - methodological aspects and effects of biofeedback-based Nintendo Wii training. Dan Med J. 2014 Jan;61(1):B4775. PMID 24393594
- [Background] Jorgensen MG, Laessoe U, Hendriksen C, Nielsen OB, Aagaard P. Efficacy of Nintendo Wii training on mechanical leg muscle function and postural balance in community-dwelling older adults: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2013 Jul;68(7):845-52. doi: 10.1093/gerona/gls222. Epub 2012 Oct 31. PMID 23114461
- [Background] King AC, Taylor CB, Haskell WL, Debusk RF. Strategies for increasing early adherence to and long-term maintenance of home-based exercise training in healthy middle-aged men and women. Am J Cardiol. 1988 Mar 1;61(8):628-32. doi: 10.1016/0002-9149(88)90778-3. PMID 3344690
- [Background] Laufer Y, Dar G, Kodesh E. Does a Wii-based exercise program enhance balance control of independently functioning older adults? A systematic review. Clin Interv Aging. 2014 Oct 23;9:1803-13. doi: 10.2147/CIA.S69673. eCollection 2014. PMID 25364238
- [Background] Palacios-Cena D, Ortiz-Gutierrez RM, Buesa-Estellez A, Galan-Del-Rio F, Cachon Perez JM, Martinez-Piedrola R, Velarde-Garcia JF, Cano-DE-LA-Cuerda R. Multiple sclerosis patients' experiences in relation to the impact of the kinect virtual home-exercise programme: a qualitative study. Eur J Phys Rehabil Med. 2016 Jun;52(3):347-55. Epub 2016 Feb 17. PMID 26883340
- [Background] Santos-Eggimann B, Cuenoud P, Spagnoli J, Junod J. Prevalence of frailty in middle-aged and older community-dwelling Europeans living in 10 countries. J Gerontol A Biol Sci Med Sci. 2009 Jun;64(6):675-81. doi: 10.1093/gerona/glp012. Epub 2009 Mar 10. PMID 19276189
- [Background] Schutzer KA, Graves BS. Barriers and motivations to exercise in older adults. Prev Med. 2004 Nov;39(5):1056-61. doi: 10.1016/j.ypmed.2004.04.003. PMID 15475041
- [Background] Walston J, McBurnie MA, Newman A, Tracy RP, Kop WJ, Hirsch CH, Gottdiener J, Fried LP; Cardiovascular Health Study. Frailty and activation of the inflammation and coagulation systems with and without clinical comorbidities: results from the Cardiovascular Health Study. Arch Intern Med. 2002 Nov 11;162(20):2333-41. doi: 10.1001/archinte.162.20.2333. PMID 12418947